CLINICAL TRIAL: NCT06217315
Title: Endometriosis and Health Care System Utilization in British Columbia
Acronym: EndoCare
Status: Active, not recruiting | Type: Observational
Sponsor: BC Women's Hospital & Health Centre (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Paul Yong, Associate Professor, BC Women's Hospital & Health Centre
Other Study IDs: H21-01699; 2023-06565 (Other Grant/Funding Number: The Swedish Research Council)
Record Dates: First submitted 2024-01-02; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention — There is no intervention.

SUMMARY:
Purpose & Background Endometriosis is a chronic inflammatory condition believed to affect 8-10% of reproductive-age women and an unmeasured number of gender-diverse people. It is a common cause of pelvic pain and infertility, is now known to be associated with other conditions such as heart disease and ovarian cancer and can have a devastating impact on a woman's ability to function and achieve their full potential. It has been shown that endometriosis and chronic pelvic pain are associated with considerable costs to the health-care system in Canada. The in-patient hospital costs for chronic pelvic pain were estimated to be $25 million/year and the total societal costs for endometriosis were estimated to be 1.8 billion/year.

Standard therapies for endometriosis and pelvic pain include pain medications, hormonal suppressive therapies, and surgery. There is a tertiary referral centre of excellence for endometriosis at BC Women's Hospital (Centre for Pelvic Pain and Endometriosis), which provides advanced surgical treatment of endometriosis and interdisciplinary care for patients with endometriosis who have developed other pain comorbidities (e.g. due to central nervous system sensitization). Central sensitization responds best to treatments targeted to the nervous system, such as Interdisciplinary care includes pain education, physiotherapy, and mindfulness-based cognitive therapies. One randomized trial has shown the benefit of an interdisciplinary approach compared to standard treatment for the management of chronic pelvic pain. At our centre, the investigators reported improvements in pain, mental health, quality-of-life, and self-reported reduction in health care utilization, after interdisciplinary care, utilizing our ongoing prospective registry. However, a formal economic analysis of health care system utilization is required to quantify savings to the health care system with an interdisciplinary approach to endometriosis.

Despite surgery being a common treatment of endometriosis, there is variability in outcome and a gap is the lack of ability to predict outcomes after endometriosis surgery. For example, utilizing self-reported outcomes from our registry, the investigators found that poorer outcome after endometriosis surgery was found in patients with evidence of pain comorbidities and central sensitization (as surgery is not a direct treatment of these factors) (in preparation). Moreover, the investigators have a biobank and have been studying biomarkers in surgically excised endometriosis tissue that may predict outcomes after surgery. These biomarkers include somatic cancer driver mutations and neuroinflammation. The investigators have preliminary data that suggests that these biomarkers may predict rates of re-operation at the centre. Beyond self-reported outcomes and re-operation at the centre, there is a need to assess health care utilization and re-operation occurring throughout the province as additional outcomes that may be associated with our clinical and biomarker predictors.

Finally, the SARS-CoV-2 (COVID-19) pandemic has had profound physical and mental health effects on populations worldwide. However, there exists limited empirical evidence focusing on the wellbeing of patients with endometriosis and/or pelvic pain during the public health crisis. Herein, the investigators propose to compare a pre-pandemic cohort to a pandemic cohort of subjects with endometriosis and/or chronic pelvic pain, again in terms of health care system utilization.

Therefore, the overall purpose of this project is to assess health care utilization patterns of patients with endometriosis in British Columbia, and to perform an economic analysis of interdisciplinary care, evaluate clinical-biomarker predictors of surgical outcome, and assess the impact of the covid pandemic. This will be achieved by linking Population Data BC datasets to our ongoing prospective registry (H16-00264) and prospective and retrospective biobanks (H14-03040, H17-00329).

DETAILED DESCRIPTION:
HYPOTHESIS Aim 1: The investigators hypothesize that health care costs for patients being cared for in our clinic will be higher in the three years preceding their time with us than the years following their discharge. The investigators hypothesize that the overall cost of the interdisciplinary clinic, including physiotherapist, counsellor and nurse salaries and administrative support, will be less than overall cost savings to the system from reduced utilization of health care resources after discharge.

Aim 2: The investigators hypothesize that comorbidities associated with central nervous system sensitization and biomarkers including somatic mutations and local neurogenesis/neuroinflammation are linked to persistent pain and disease recurrence after endometriosis surgery, which results in increased risk of re-operation and health care utilization after surgery.

Aim 3: The pandemic cohort will have increased health care system utilization, and also poorer health system outcomes after care the centre.

Aim 4: People with endometriosis, utilizing different case definitions, will experience higher health care use and worse pregnancy outcomes, compared to people without endometriosis.

ELIGIBILITY:
The cohort will consist of all females in British Columbia between January 1st 2000 and December 31st 2021 as identified by the Consolidation File Dataset available by Population Health Data BC.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The cohort will consist of all females in British Columbia between January 1st 2000 and December 31st 2021 as identified by the Consolidation File Dataset available by Population Health Data BC.
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Economic Impact | Jan 1st 2000 - Dec 31st 2021
  To assess the cost-effectiveness of an interdisciplinary model of care for endometriosis by measuring the cost of healthcare services as determined by BC Medical Service Plan billing codes.
Prediction Model | Jan 1st 2000 - Dec 31st 2021
  To identify clinical and biomarker predictors and quality of life after surgery as measured by the Endometriosis Health Profile (EHP-30).
Covid pre-post outcomes | Jan 1st 2000 - Dec 31st 2021
  To determine the impact of the COVID-19 pandemic on health care system utilization of patients with endometriosis by measuring clinical biomarkers, KRAS mutations and quality of life outcomes (EHP-30, GAD-7, PHQ-9, Central Sensitization Inventory CSI) before and after the pandemic.
Impact of Health Care Utilization | Jan 1st 2000 - Dec 31st 2021
  To understand the overall impact of endometriosis on health care use, including with respect to surgical and pregnancy outcomes as measured by number of surgical operations, medication use and live birth rates.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Yong, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital + Health Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
Metadata can be shared with other researchers. Raw data is restricted.